CLINICAL TRIAL: NCT00235391
Title: A Study to Provide Expanded Access of (Exjade®) Deferasirox to Patients With Congenital Disorders of Red Blood Cells and Chronic Iron Overload From Blood Transfusions Who Cannot Adequately be Treated With Other Locally Approved Iron Chelators
Brief Title: Expanded Access of Deferasirox to Patients With Congenital Disorders of Red Blood Cells and Chronic Iron Overload
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670A2203
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Results first posted 2011-05-02 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2011-06

CONDITIONS: Thalassemia; Sickle Cell Disease; Diamond Blackfan Anemia; Myelofibrosis
Keywords: Deferasirox; Congenital Anemias; Anemias; Red Blood Cell Disorders; Chronic Iron Overload; Transfusional Iron Overload; Iron Chelators; Oral Iron Chelators; Thalassemia; Sickle Cell Disease; Diamond Blackfan Anemia; Myelofibrosis; ICL670A
MeSH Terms: conditions — Thalassemia; Anemia, Sickle Cell; Anemia, Diamond-Blackfan; Primary Myelofibrosis; Anemia | interventions — Deferasirox

ARMS (1):
- Deferasirox (Experimental): Deferasirox was administered orally once a day, 30 minutes prior to breakfast. Dosage was based on participant's body weight. Starting dose was determined by the frequency of blood transfusions and recommended initial daily dose of deferasirox is 20 mg/kg body weight for patients receiving blood transfusion, 10 mg/kg for patients receiving less frequent transfusion/exchange transfusion and 30 mg/kg for patients receiving more frequent blood transfusions.
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferasirox — 125 mg, 250 mg and 500 mg tablets. Dosage was calculated based on participant's body weight. Tablets were dispersed in water, orange or apple juice and taken orally once a day.

SUMMARY:
This is an open-label, non-randomized, multi-center trial designed to provide expanded access of deferasirox to patients with congenital disorders of red blood cells and chronic iron overload from blood transfusions who cannot adequately be treated with locally approved iron chelators.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients greater than or equal to 2 years of age
* Documented congenital disorder of red blood cells (e.g., β-thalassemia major, sickle cell anemia, diamond-blackfan anemia) requiring ongoing blood transfusions
* Cannot be adequately treated with a locally approved iron chelator due to one of the following reasons:

  * Documented non-compliance, defined as having taken less than 50% of the prescribed chelation therapy doses in the 12 months prior to study entry
  * Contraindications, unacceptable toxicities and/or documented poor response to locally approved iron chelators despite proper compliance
* History of at least 20 blood transfusions (equivalent to 100 mL/kg of packed red blood cells (PRBC])
* Serum ferritin value greater than or equal to 1000 µg/L
* Ability to comply with all study-related procedures, medications, and evaluations

Exclusion Criteria:

* Ongoing treatment with another iron chelator (Any other iron chelation therapy must be discontinued at least 24 hours prior to study entry.)
* Patients who meet the eligibility criteria for any other ongoing Novartis sponsored clinical study protocol with deferasirox and who have geographic access to these sites
* Patients unable to tolerate (or who have unacceptable toxicities to) prior treatment with deferasirox
* Serum creatinine above the upper limit of normal at screening.
* Patients with ALT ≥ 500 U/L at screening.
* Evidence of chelation-related cataracts or hearing loss within 4 weeks prior to baseline
* Pregnancy (as indicated by serum β-HCG pregnancy test at screening for all female patients with the potential to become pregnant) and patients who are breastfeeding
* Patients treated with systemic investigational drug within 4 weeks prior to or with topical investigational drug within 7 days prior to the baseline visit

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1683 (Actual)
Dates: Start 2005-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (141):
- United States (27):
  - Arkansas Children's Hospital, UAMS College of Medicine, Little Rock, Arkansas
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Children's Hospital of Orange County, Orange, California
  - Children's Hospital and Health Center of San Diego, San Diego, California
  - Stanford University, Stanford, California
  - Alfred I. Dupong Hospital for Children, Wilmington, Delaware
  - Osler Medical, Inc., Melbourne, Florida
  - Hematalogy Oncology Associates, Pensacola, Florida
  - Tampa Children's Hospital at St. Joseph's Hospital, Tampa, Florida
  - James A. Haley Veterans Hospital, Tampa, Florida
  - Backus Children's Hospital, Memorial Health University Medical Center, Savannah, Georgia
  - Hematalogy Oncology Clinic, Baton Rouge, Louisiana
  - Borgess Hospital, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - The Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Schneider Children's Hospital, New Hyde Park, New York
  - PCTI, Columbus, Ohio
  - The Children's Medical Center of Dayton, Dayton, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospitals of Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Children's Hospital of the Kings Daughters, Norfolk, Virginia
  - VCU Pediatric Hematology/Oncology, Richmond, Virginia
  - University of Washington Seattle Cancer Care Alliance, Seattle, Washington
- Belgium (4):
  - Ziekenhuisnetwerk Antwerpen-AZ Middelheim, Antwerp
  - Centre Hospitalier Notre Dame et Reine, Charleroi
  - CHR de la Citadelle, Liège
  - Centre Hospitalier Chretien-Clinique Saint-Joseph, Montegnée
- Canada (9):
  - The Ottawa Hospital-General Campus, Ottawa, Ontario
  - University of Alberta, Edmonton
  - CHUM-Hopital-Notre-Dame, Montreal
  - MUHC- Montreal Children's Hospital, Montreal
  - MUHC- Royal Victoria Hospital, Montreal
  - Hopital de l'Enfant-Jesus, Québec
  - The Hospital for Sick Children,, Toronto
  - Toronto General Hospital-Hemoglobinopathy, Toronto
  - Burrard Medical Building, Vancouver
- Germany (9):
  - Charite-Universitatsmedizin Berlin, Berlin
  - Universitatsklinikum Koln, Cologne
  - Universitaetsklinik Dusseldorf, Düsseldorf
  - Johann Wolfgang von Goethe Universitat, Frankfurt am Main
  - Georg-August-Universitat Gottingen, Göttingen
  - Universitatskrankenhaus Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum Stuttgart Bismarckstrasse 8, Stuttgart
  - Universitatsklinikum Ulm, Ulm
- Greece (18):
  - Agia Sofia Hospital of Athens, Athens
  - General Hospital of Athens, Athens
  - Ippokration Hospital of Athens, Athens
  - General Hospital of Athens, Corfu
  - General Hospital of Korinthos, Corinth
  - General Hospital of Heraklion Benizeleio-Pananeio, Heraklion
  - University Hospital of Ioannina, Ioannina
  - General Hospital of Kalamata, Kalamata
  - Agia Sofia Hospital of Athens, Karditsa
  - General Hospital of Karditsa, Karditsa
  - General Hospital of Larisa Tsakalof 1, Larissa
  - General Hospital of Mytilini Vostaneio, Mytilene
  - General State Hospital of Nikaia St. Panteleimon, Nikaia
  - University Hospital of Patras, Pátrai
  - General Hospital of Thessaloniki Agios Pavlos, Thessaloniki
  - General Hospital Thessalonikis Hippokratio, Thessaloniki
  - General Hospital of Volos, Volos
  - General Hospital of Xanthi, Xánthi
- Italy (36):
  - Presidio Ospedale Muscatello, Augusta
  - A.O. Ospedale Policlinico Consorziale di Bari, Bari
  - Presidio Ospedaliero Antonio Perrino, Brindisi
  - Ospedale Regionale Microcitemie, Cagliari
  - Ospedale Di Venere, Carbonara di Bari
  - Azienda Ospedali Vittorio Emanuele, Ferrarotto e San Bambino, Catania
  - Presidio Ospedaliero S. Bambino, Catania
  - PresidioOspedaliero S. Luigi Curro, Catania
  - Azienda Ospedaliera Pugliese Cicaccio, Catanzaro
  - Ospedale Civile dell'Annunziata, Cosenza
  - Ospedale San Giuseppe, Empoli
  - Azienda Ospedaliera Universitaria di Ferrara, Ferrara
  - Azienda Ospedaliera A. Meyer, Florence
  - E.O. Ospedali Galliera, Genova
  - Ospedale Regionale Microcitemie, Itala
  - Ospedale Madonna delle Grazie, Matera
  - Az. Ospedaliera Universitaria Policlinico G. Martino, Messina
  - Fondazione Ospedale, Milan
  - Azienda Ospedaliero-Universitaria di Modena, Modena
  - AORN A. Cardarelli, Napoli
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliera V. Cervello, Palermo
  - Azienda Ospedaliera Villa Sofia-CTO, Palermo
  - Presidio Ospedaliero Giovanni di Cristina, Palermo
  - IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliera San Salvatore, Pesaro
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Ospedaliera Civile- Maria Paterno, Ragusa
  - Azienda Ospedaliera Bianchi-Melacrino-Morelli, Reggio Calabria
  - Ospedale S. Eugenio, Roma
  - Ospedale nostra Signora di Bonaria, San Gavino Monreale- CA
  - Presidio Ospedaliero di Sassari-Ospedale SS, Sassari
  - Azienda Ospedaliera Ospedali Civili Riuniti di Sciacca, Sciacca
  - Ospedale Umberto I, Talassemie
  - Presidio Ospedaliero Centrale, Taranto
  - Ospedale Infantile Regina Margherita, Torino
- Netherlands (5):
  - AMC, Amsterdam
  - Catharina-ziekenhuis, Eindhoven
  - Erasmus MC, Rotterdam
  - Erasmus Medisch Centrum, locatie Sophia, Rotterdam
  - Haga Ziekenhuis, The Hague
- Spain (11):
  - Hospital de Torrecardenas, Almería
  - Hospital Infanta Cristina, Badajoz
  - Hospital Cruces, Barakaldo
  - Hospital Puerta del Mar, Cadiz
  - Hospital De Gran Canaria, Canara
  - Hospital Universitario La Paz, Madrid
  - Althaia : Xarxa Assistencial de Manresa, Manresa
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Virgen de la Salud, Toledo
  - Hospital Universitario La Fe, Valencia
  - Hospital Xeral de Vigo, Vigo
- Taiwan (5):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Mackay Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Chang Gung Children's Hospital, Taoyuan District
  - Tao-yuan General Hospital, Tau-Yuan County
- Thailand (4):
  - Phramongkutklao Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Songklanagarind Hospital, Bangkok
  - Srinagarind Hospital, Khon Kaen
- Turkey (Türkiye) (8):
  - Cukurova Universitesi, Adana
  - Hacettepe Universitesi, Ankara
  - Akdeniz Universitesi, Antalya
  - Gaziantep Universitesi, Gaziantep
  - Suleyman Demirel, Isparta
  - Istanbul Universitesi, Istanbul
  - Ege Universitesi Tip Fakultesi, Izmir
  - Erciyes Universitesi, Kayseri
- United Kingdom (5):
  - Evelina Hospital St. Thomas' Hospital, London
  - North Middlesex University Hospital, London
  - The Royal Hospital London, London
  - Whittington Hospital, London
  - St. George's Hospital, Tooting

REFERENCES:
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.novartisclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- 2 to < 6 Years; 6 to < 12 Years; 12 to < 16 Years; 16 to < 50 Years; 50 to < 65 Years; ≥ 65 Years: Deferasirox was administered orally once a day, 30 minutes prior to breakfast. Dosage was based on participant's body weight. Tablets were dispersed in water, orange or apple juice.
Period: Overall Study
Arm/Group | 2 to < 6 Years | 6 to < 12 Years | 12 to < 16 Years | 16 to < 50 Years | 50 to < 65 Years | ≥ 65 Years
Started | 97 | 200 | 172 | 1164 | 43 | 7
Deferasirox Treatment | 97 | 200 | 172 | 1164 | 43 | 7
Completed | 85 | 182 | 148 | 944 | 31 | 3
Not Completed | 12 | 18 | 24 | 220 | 12 | 4
Not completed — Adverse Event | 4 | 5 | 10 | 72 | 5 | 2
Not completed — Abnormal laboratory value(s) | 3 | 5 | 4 | 27 | 1 | 2
Not completed — Unsatisfactory therapeutic effect | 0 | 2 | 2 | 17 | 0 | 0
Not completed — Condition no longer requires treatment | 3 | 0 | 0 | 11 | 1 | 0
Not completed — Protocol deviation | 0 | 0 | 1 | 11 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 3 | 61 | 5 | 0
Not completed — Lost to Follow-up | 0 | 3 | 3 | 16 | 0 | 0
Not completed — Administrative problems | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2 to < 6 Years | 6 to < 12 Years | 12 to < 16 Years | 16 to < 50 Years | 50 to < 65 Years | ≥ 65 Years | Total
Number analyzed (Participants) | 97 | 200 | 172 | 1164 | 43 | 7 | 1683
Age Continuous [Mean (Standard Deviation); unit: years] | 3.48 (1.13) | 8.52 (1.64) | 13.48 (1.20) | 28.91 (8.06) | 54.58 (3.92) | 70.14 (3.98) | 24.27 (12.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 101 | 81 | 633 | 32 | 5 | 896
  Male | 53 | 99 | 91 | 531 | 11 | 2 | 787
Baseline Disease Characteristics [Number; unit: participants] — The number of participants with each disease category.
  participants
    Beta-Thalassemia Major | 74 | 118 | 114 | 905 | 10 | 0 | 1221
    Beta-Thalassemia Intermedia | 1 | 22 | 16 | 94 | 20 | 3 | 156
    Sickle Cell Disease | 8 | 41 | 31 | 93 | 2 | 1 | 176
    Diamond-Blackfan Anemia | 4 | 7 | 8 | 24 | 0 | 0 | 43
    Other Diseases | 10 | 12 | 3 | 48 | 11 | 3 | 87
Prior Chelation Drug Therapy [Number; unit: participants] — The number of participants for each chelation drug category.
  participants
    Deferoxamine | 80 | 167 | 137 | 745 | 31 | 5 | 1165
    Deferiprone | 1 | 8 | 11 | 146 | 6 | 1 | 173
    Deferoxamine and Deferiprone | 2 | 16 | 21 | 269 | 6 | 0 | 314
    Other Chelation Drug | 6 | 6 | 3 | 4 | 0 | 0 | 19
    Prior Chelatation Drug Information Missing | 8 | 3 | 0 | 0 | 0 | 1 | 12
Reason for inadequate prior chelation therapy [Number; unit: participants] — The number of participants for each reason for inadequate prior chelation therapy category.
  participants
    Therapy non-compliance | 57 | 125 | 106 | 659 | 25 | 2 | 974
    Therapy contraindication | 1 | 7 | 6 | 29 | 1 | 1 | 45
    Therapy unacceptable toxicity | 11 | 29 | 22 | 131 | 6 | 1 | 200
    Therapy poor response | 20 | 34 | 38 | 267 | 8 | 0 | 367
    Therapy unacceptable discomfort | 2 | 2 | 0 | 78 | 3 | 2 | 87
    Reason for inadequate therapy information missing | 6 | 3 | 0 | 0 | 0 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Safety Profile of Deferasirox Based Upon Drug Administration and Reporting of Serious Adverse Events
Description: Safety as assessed by the number of participants with death, serious adverse events (SAE), and/or Adverse Events (AEs) leading to study drug interruption or discontinuation. Note: only treatment emergent AEs are summarized.
Time Frame: Baseline to end of study (Median exposure time to drug was approximately 30 weeks; Maximum exposure was 104 weeks)
Population: The safety population, comprising all participants who received at least one dose of deferasirox during the study, was used in the analyses.
Measure: Number; unit: Participants
Arm/Group | 2 to < 6 Years | 6 to < 12 Years | 12 to < 16 Years | 16 to < 50 Years | 50 to < 65 Years | ≥ 65 Years
Number analyzed (Participants) | 97 | 200 | 172 | 1164 | 43 | 7
Participants
  Number of deaths | 0 | 0 | 1 | 4 | 0 | 0
  Non-fatal SAEs | 10 | 22 | 27 | 129 | 4 | 2
  AEs leading to discontinuation | 4 | 5 | 10 | 75 | 5 | 2
  AEs leading dose adjustment/temporary interruption | 15 | 31 | 28 | 209 | 11 | 2

2. Secondary Outcome: The Change in Serum Ferritin Values From Baseline Through Completion of the Study
Description: The number of participants with Improvement, No Change or Worsening in Serum ferritin category levels at the end of the study compared to baseline. Serum ferritin levels in µg/L were divided into to 6 categories: (<1000), (1000-<2500), (2500-<4000), (4000-<5500), (5500-<7000) and (>=7000). Improvement was defined as a shift to a lower category at the end of study compared to the category at baseline. Worsening was defined as a shift to a higher category at the end of the study compared to the category at baseline. No change was no change in category at end of study from baseline.
Time Frame: Baseline to end of study (Median exposure time to drug was approximately 30 weeks; Maximum exposure was 104 weeks)
Population: Safety population defined as all participants who received at least one dose of study drug. This analysis did not include participants with unknown status at baseline and/or at the end of the study.
Measure: Number; unit: Participants
Arm/Group | 2 to < 6 Years | 6 to < 12 Years | 12 to < 16 Years | 16 to < 50 Years | 50 to < 65 Years | ≥ 65 Years
Number analyzed (Participants) | 97 | 200 | 172 | 1164 | 43 | 7
Participants
  Improvement | 17 | 27 | 26 | 206 | 4 | 2
  No Change | 63 | 106 | 87 | 570 | 31 | 3
  Worsening | 16 | 63 | 55 | 341 | 7 | 1

ADVERSE EVENTS:
Groups:
- All Participants: Deferasirox was administered orally once a day, 30 minutes prior to breakfast. Dosage was based on participant's body weight. Tablets were dispersed in water, orange or apple juice.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 194/1683
Other Adverse Events (participants affected / at risk) | 85/1683
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=1683)
Acute chest syndrome (Blood and lymphatic system disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 2
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 2
Coombs positive haemolytic anaemia (Blood and lymphatic system disorders) | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1
Hypersplenism (Blood and lymphatic system disorders) | 3
Intravascular haemolysis (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Pancytopenia (Blood and lymphatic system disorders) | 1
Reticulocytopenia (Blood and lymphatic system disorders) | 1
Splenomegaly (Blood and lymphatic system disorders) | 4
Arrhythmia (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 6
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 2
Congestive cardiomyopathy (Cardiac disorders) | 1
Myopericarditis (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ventricular dysfunction (Cardiac disorders) | 1
Hip dysplasia (Congenital, familial and genetic disorders) | 1
Sickle cell anaemia (Congenital, familial and genetic disorders) | 2
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 27
Thalassaemia (Congenital, familial and genetic disorders) | 1
Thalassaemia beta (Congenital, familial and genetic disorders) | 2
Deafness unilateral (Ear and labyrinth disorders) | 1
Middle ear effusion (Ear and labyrinth disorders) | 1
Retinopathy (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Crohn's disease (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 4
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Catheter thrombosis (General disorders) | 1
Death (General disorders) | 1
Local swelling (General disorders) | 1
Malaise (General disorders) | 3
Non-cardiac chest pain (General disorders) | 5
Pain (General disorders) | 3
Pyrexia (General disorders) | 9
Biliary colic (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 6
Hepatitis (Hepatobiliary disorders) | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Abdominal infection (Infections and infestations) | 1
Acute tonsillitis (Infections and infestations) | 2
Appendicitis (Infections and infestations) | 1
Bacterial infection (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 2
Bronchopneumonia (Infections and infestations) | 1
Catheter related infection (Infections and infestations) | 1
Catheter site infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 2
Diarrhoea infectious (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Epstein-Barr virus infection (Infections and infestations) | 3
Escherichia bacteraemia (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 3
Gastrointestinal infection (Infections and infestations) | 1
Hepatitis C (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Necrotising fasciitis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 2
Otitis media acute (Infections and infestations) | 1
Parvovirus infection (Infections and infestations) | 1
Perianal abscess (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 4
Pyelonephritis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 5
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 2
Forearm fracture (Injury, poisoning and procedural complications) | 1
Haemolytic transfusion reaction (Injury, poisoning and procedural complications) | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 2
Spinal fracture (Injury, poisoning and procedural complications) | 1
Suture rupture (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Blood calcium increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Cardiovascular evaluation (Investigations) | 1
Protein urine present (Investigations) | 1
Serum ferritin increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Benign neoplasm of thymus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic neoplasm malignant recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Convulsion (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Migraine (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 5
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Calculus ureteric (Renal and urinary disorders) | 1
Nephrotic syndrome (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 2
Urethral stenosis (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1
Uterine disorder (Reproductive system and breast disorders) | 1
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Swelling face (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Uterine dilation and curettage (Surgical and medical procedures) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=1683)
Rash (Skin and subcutaneous tissue disorders) | 85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.